CLINICAL TRIAL: NCT06754904
Title: OMIT Trial: Omitting Therapeutic Lymph Node Dissection in Patients With Stage IIIB/C Melanoma and Major Pathological Response in the Index Lymph Node After Neoadjudvant Immunotherapy
Brief Title: Omitting Therapeutic Lymph Node Dissection in Patients With Melanoma (Stage 3) and Major Pathological Response in the Index Lymph Node
Acronym: OMIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: D.J. (Dirk) Grünhagen (Other)
Responsible Party: Sponsor-Investigator, D.J. (Dirk) Grünhagen, Associate professor, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL88017.078.24; NL88017.078.24 (Registry Identifier: CCMO)
Record Dates: First submitted 2024-12-13; First posted 2025-01-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Melanoma, Skin
Keywords: Neoadjuvant; Ipilimumab; Nivolumab; Immunotherapy; Index node; Therapeutic lymph node dissection; Omitting
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Omitting TLND in patients who achieve an MPR in the ILN following neoadjuvant ipilimumab and nivolumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omitting TLND (Experimental): Omitting TLND in patients who achieve an MPR in the ILN following neoadjuvant ipilimumab and nivolumab.
  Interventions: Procedure: Omitting TLND; Procedure: Index node procedure

INTERVENTIONS:
Procedure: Omitting TLND — Omitting TLND in patients who achieve an MPR in the index node following neoadjuvant ipilimumab and nivolumab.
Procedure: Index node procedure — Index node procedure

SUMMARY:
Rationale: The randomized trial NADINA has demonstrated that neoadjuvant treatment with nivolumab with ipilimumab improves event-free survival (EFS) in patients with macroscopic resectable stage III melanoma. In this study, therapeutic lymph node dissection (TLND) was standard of care, showing that patients achieving a major pathological response (MPR, i.e., ≤10% residual viable tumor bed) have an excellent outcome (EFS and Distant Metastasis Free Survival (DMFS)). The PRADO trial indicated that the MPR definition can also be revealed from a surrogate lymph node response, the index lymph node (ILN), allowing sparing the extensive surgery in MPR patients. In these MPR patients the DMFS was 100% after 1 year and 98% after 2 years, and recurrence-free survival (RFS) was 95% after 1 year and 93% after 2 years. Given that TLND is associated with morbidity and has a significant impact on health-related quality of life (HR-QoL) and healthcare costs, this study aims to prospectively investigate the safety of omitting TLND in patients who have an MPR within the ILN after neoadjuvant immunotherapy.

Objectives: To investigate whether TLND can be safely omitted in patients with macroscopic resectable stage III (B/C/D) melanoma achieving an MPR within the ILN upon neoadjuvant treatment with immune checkpoint inhibitors (ipilimumab and nivolumab).

Study design: This study is a prospective, single-arm phase 2 nationwide multicenter trial.

Study population:

Inclusion criteria for study participants are as follows:

* Patients must be eligible for neoadjuvant treatment
* Patients must have a histologically confirmed diagnosis of macroscopic resectable stage III melanoma (stage III B/C/D) with one or more macroscopic lymph node metastasis
* The patient must have a measurable tumor burden that qualifies (according to clinical practice) for neoadjuvant therapy

Intervention: Omitting TLND in patients who achieve an MPR in the ILN following neoadjuvant ipilimumab and nivolumab.

Main study endpoints: The two coprimary endpoints are 2-year Local Recurrence Free Survival (LRFS) and 2-year DMFS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be eligible for neoadjuvant treatment (ipilimumab and nivolumab)
* Patients must be 16 years of age or older.
* Patients must have a histologically confirmed diagnosis of macroscopic resectable stage III melanoma (stage III B/C/D) with one or more macroscopic lymph node metastase defined as either one:
* a palpable node, confirmed as melanoma by pathology; a non-palpable but enlarged lymph node according to RECISTv1.1 (at least 15 mm in short axis), confirmed as melanoma by pathology;
* a PET scan positive lymph node of any size confirmed as melanoma by pathology;
* The patient must have a measurable tumor burden that qualifies (according to clinical practice) for neoadjuvant therapy with immune checkpoint inhibitors
* Patients in whom ILN marking is feasible
* Written informed consent

Exclusion Criteria:

* Uveal/ocular or mucosal melanoma
* WHO performance status of two or more
* In-transit metastases only (without cytological or histological proven lymph node involvement)
* Prior targeted therapy targeting BRAF and/or MEK for melanoma
* Prior immunotherapy targeting CTLA-4, PD-1 or PD-L1 for melanoma
* Patients with (history of) distant metastasis (stage IV melanoma)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Local Recurrence Free Survival (LRFS) | 2 years after inclusion
  LRFS, as defined as time from removal of the index lymph node (ILN) until local (in basin) recurrence in the MPR group. Accepting a local relapse of 20%.
Distant Metastasis Free Survival (DMFS) | 2 years after inclusion
  DMFS assessed in the MPR group, as defined as time from the start of neoadjuvant immunotherapy, nivolumab with ipilimumab, until the first occurrence of distant metastasis. Accepting DMFS 3% lower than the 2 years DMFS of the NADINA trial

SECONDARY OUTCOMES:
Evaluation of health-related quality of life (HRQoL), EORTC QLQ C30 | 3 years after inclusion
  Description of the changes in HR-QoL scores from baseline to follow-up visits, measured by validated questionnaires using EORTC Quality of Life Questionnaire-core 30 (EORTC QLQ C30). The EORTC QLQ C30 is scored on 4 point Likert-scales: "Not at all", "A little", "Quite a bit", and "Very much."
Evaluation of health-related quality of life (HRQoL), FACT-M | 3 years after inclusion
  Description of the changes in HR-QoL scores from baseline to follow-up visits, measured by validated questionnaires using Melanoma Surgery Specific subscale of the FACT-M. The FACT-M is scored on a 5 point Likert-scale: "Not at all", "A little bit", "Somewhat", "Quite a bit", and "Very much."
Description of the pathological response rates in the ILN | 1 year after inclusion
  The pathologic response rate is categorized into pathologic complete response (pCR), near-pCR, major pathologic response (MPR), pathologic partial response (pPR), pathologic no response (pNR), according to International Neoadjuvant Melanoma Consortium (INMC) criteria.
Evaluation of the surgical morbidity, CTCAE v5 | 2 year after inclusion
  Description of the incidence and severity of post-surgical complications according to CTCAE v5
Evaluation of the surgical morbidity, Clavien Dindo | 2 year after inclusion
  Description of the incidence and severity of post-surgical complications according to Clavien Dindo
Radiological evaluation of the index lymph node | 1 year after inclusion
  Calculate Concordance rates between radiological and pathological response (pCR, pPR, pNR) in the ILN
Proportion of patients undergoing therapeutic lymph node dissection (TLND) | 5 years after inclusion
  Description of the proportion of patients undergoing TLND stratified by MPR and non-MPR status
Melanoma specific survival | 5 years after inclusion
  Description of the Melanoma specific survival, as calculated time from the date of start of neoadjuvant therapy to the date of death due to melanoma
Overall survival | 5 years after inclusion
  Description of the overall survival, as calculated time from the date of start of neoadjuvant therapy to the date of death due to melanoma or any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
We have decided not to share de-identified individual participant data, as the dataset is intended for exclusive use by the primary research group. Sharing the data with researchers outside of this group is not aligned with the original goals and agreements of the study.
  Should there be a need for collaboration or data sharing in the future, we will evaluate this in consultation with the relevant parties.

REFERENCES:
- [Background] Blank CU, Lucas MW, Scolyer RA, van de Wiel BA, Menzies AM, Lopez-Yurda M, Hoeijmakers LL, Saw RPM, Lijnsvelt JM, Maher NG, Pulleman SM, Gonzalez M, Torres Acosta A, van Houdt WJ, Lo SN, Kuijpers AMJ, Spillane A, Klop WMC, Pennington TE, Zuur CL, Shannon KF, Seinstra BA, Rawson RV, Haanen JBAG, Ch'ng S, Naipal KAT, Stretch J, van Thienen JV, Rtshiladze MA, Wilgenhof S, Kapoor R, Meerveld-Eggink A, Grijpink-Ongering LG, van Akkooi ACJ, Reijers ILM, Gyorki DE, Grunhagen DJ, Speetjens FM, Vliek SB, Placzke J, Spain L, Stassen RC, Amini-Adle M, Lebbe C, Faries MB, Robert C, Ascierto PA, van Rijn R, van den Berkmortel FWPJ, Piersma D, van der Westhuizen A, Vreugdenhil G, Aarts MJB, Stevense-den Boer MAM, Atkinson V, Khattak M, Andrews MC, van den Eertwegh AJM, Boers-Sonderen MJ, Hospers GAP, Carlino MS, de Groot JB, Kapiteijn E, Suijkerbuijk KPM, Rutkowski P, Sandhu S, van der Veldt AAM, Long GV. Neoadjuvant Nivolumab and Ipilimumab in Resectable Stage III Melanoma. N Engl J Med. 2024 Nov 7;391(18):1696-1708. doi: 10.1056/NEJMoa2402604. Epub 2024 Jun 2. PMID 38828984
- [Background] Reijers ILM, Menzies AM, van Akkooi ACJ, Versluis JM, van den Heuvel NMJ, Saw RPM, Pennington TE, Kapiteijn E, van der Veldt AAM, Suijkerbuijk KPM, Hospers GAP, Rozeman EA, Klop WMC, van Houdt WJ, Sikorska K, van der Hage JA, Grunhagen DJ, Wouters MW, Witkamp AJ, Zuur CL, Lijnsvelt JM, Torres Acosta A, Grijpink-Ongering LG, Gonzalez M, Jozwiak K, Bierman C, Shannon KF, Ch'ng S, Colebatch AJ, Spillane AJ, Haanen JBAG, Rawson RV, van de Wiel BA, van de Poll-Franse LV, Scolyer RA, Boekhout AH, Long GV, Blank CU. Personalized response-directed surgery and adjuvant therapy after neoadjuvant ipilimumab and nivolumab in high-risk stage III melanoma: the PRADO trial. Nat Med. 2022 Jun;28(6):1178-1188. doi: 10.1038/s41591-022-01851-x. Epub 2022 Jun 5. PMID 35661157